CLINICAL TRIAL: NCT03243695
Title: Implant Failure When Using Angled Versus Straight Abutments in Immediately Placed and Restored Implants in the Esthetic Zone Using Computer Aided Surgical Guides:A Randomized Clinical Trial
Brief Title: Influence of Abutment Angulation on Implant Failure in Immediately Placed and Restored Implants in the Esthetic Zone Using Computer Aided Surgical Guides: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Huda Fakhry Fouad, Assistant lecturer Prosthodontic department Faculty of Dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Prosth department
Record Dates: First submitted 2017-08-04; First posted 2017-08-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Immediate Dental Implants
Keywords: immediate implants, implant failure, angled abutments

STUDY DESIGN:
Who Masked: Participant
Masking Description: due to the nature of the study only the participant could be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Angled abutment (Experimental): According to the allocation, the experimental group will receive an angled abutment on the immediately placed implant. A vaccum stent will be used to fabricate a temporary crown using tooth colored auto-polymerizing resin(structur 2 SC/ QM , VOCO GmbH, Germany)
  Interventions: Other: Angled Abutment
- Straight abutment (Active Comparator): According to the allocation, the control group will receive on the immediately placed implant a Straight zero degree abutment . A vaccum stent will be used to fabricate a temporary crown using tooth colored auto-polymerizing resin(structur 2 SC/ QM , VOCO GmbH, Germany)
  Interventions: Other: straight abutment

INTERVENTIONS:
Other: Angled Abutment — virtual implants will be placed on a planning software allowing abutments to be placed at an angle to the implant. Teeth will be extracted at the surgery using periotome and implants will be placed using computer aided surgical guide. The angled abutment will be placed and a temporary crown material will be fabricated.
  Arms: Angled abutment
Other: straight abutment — virtual implants will be placed on a planning software allowing abutments to be placed at straight to the implant. Teeth will be extracted at the surgery using periotome and implants will be placed using computer aided surgical guide. The straight abutment will be placed and a temporary crown material will be fabricated.
  Arms: Straight abutment

SUMMARY:
patients with fractured teeth in the esthetic area requiring immediate restoration will be recruited to the study. Immediate implants will be placed and patients will be restored either with straight or angled abutments. Implant failure will be measured.

DETAILED DESCRIPTION:
A: General operative procedures:

The study will be explained in details to the eligible participants with all possible alternative treatment options and possible risk.

If a patient accepts the treatment, informed consent will be signed. Standard extra oral and intraoral examination will be carried out. Diagnostic charts will be filled including medical and past dental history.

The patient will choose a sealed envelope to determine the allocation group. Preliminary impressions will be taken. The tooth to be extracted will be trimmed from the cast and an ideal wax up will be done.

A hard vacuum stent 2 mm thickness will be constructed over the cast with the wax up for fabrication of the temporary crown later.

The patient will be imaged a cone beam computerized topography (CBCT). The acquired DICOM image will be assessed on blue sky software ®. All the cases must have adequate buccolingual bone, if not the patient will be excluded from the study.

The co-supervisor (MW) will inform the principle investigator (HF) with the allocation group.

The principle investigator (HF) will plan the case. The implants will be planned apical to socket depth to engage apical bone for better primary stability. Final implant position 3 dimensionally will be according to allocation group to allow for placement of either straight or angled abutment.

The guide will be exported from the software and printed.

Intra operative procedures:

Patients will administrate a prophylactic antibiotic 3 days ahead the surgery. The procedure will be carried out under local anesthesia under sterile conditions.

The remaining tooth will be extracted atraumatically using periotome for better bone preservation.

After tooth extraction, the socket will be curettaged and irrigated with copious saline till fresh bleeding from the socket is observed.

Surgical guide will be placed and checked for stability and drilling will be performed following instructions.

Before implant insertion, the prepared osteotomy will be lavaged thoroughly to remove any drill debris from the socket.

The implant will be placed and the insertion torque will be checked using manual torque wrench. Implants with insertion torque less than 35Ncm will not be loaded and will be excluded from the study.

Periapical radiographs will be taken to ensure proper seating of the implant. The abutment, whether straight or angled according to the allocation group, will be attached to the implant fixture.

The vacuum stent will be used to perform the temporary crown using autopolymerizing resin. The crown will be checked to be out of occlusion in centric and eccentric occlusion to avoid any premature contact and subsequent overloading. Then the crown will be cemented and excess cement will be removed using dental floss.

The patient will be called for follow up after 1 week for the first 3 weeks then at 1 month and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with teeth or remaining roots indicated for extraction in the esthetic zone and eligible for immediate implant placement Sufficient bone labially (at least 1.5-2 mm) assessed after cone beam computer tomography (CBCT) scan Presence of adequate mesio distal length between the adjacent natural teeth (at least 7 mm), measured on the study cast Presence of adjacent natural teeth to the tooth/teeth to be extracted

Exclusion Criteria:

* Presence of active signs or symptoms of acute infection in the tooth or the remaining root Heavy smokers (more than 2 packs per day) Parafunctional habits (clenching or bruxism) diagnosed by history taking and observation of the occlusal surface of the posterior teeth for wear facets Patients with poor oral hygiene Pregnant women Any systemic condition that may interfere with osseointegration (as uncontrolled diabetes, recent head and neck radiation) Severe overeruption of the opposing teeth to avoid any premature contact with the temporary crown during the osseointegration period.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Implant failure | 3 months interval
  clinical observation

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Araújo, M.G. et al., 2005. Ridge alterations following implant placement in fresh extraction sockets: an experimental study in the dog. Journal of clinical periodontology, 32(6), pp.645-52. Brosh, T., Pilo, R. & Sudai, D., 1998. The influence of abutment angulation on strains and stresses along the implant/bone interface: comparison between two experimental techniques. The Journal of prosthetic dentistry, 79(3), pp.328-34. Chrcanovic, B.R., Albrektsson, T. & Wennerberg, A., 2015. Tilted versus axially placed dental implants: a meta-analysis. Journal of dentistry, 43(2), pp.149-70. Del Fabbro, M. et al., 2015. Immediate loading of postextraction implants in the esthetic area: systematic review of the literature. Clinical implant dentistry and related research, 17(1), pp.52-70.